CLINICAL TRIAL: NCT01822236
Title: Effectiveness of a Craniosacral Therapy Program on Disability, Quality of Life, Autonomic Nervous System and Oxidative Stress Indicators in Chronic Low Back Pain: a Randomized Controlled Clinical Trial
Brief Title: Craniosacral Therapy to Treat Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Collaborators: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Adelaida María Castro-Sánchez, PhD (Lecturer), Universidad de Almeria
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: UAL-123
Record Dates: First submitted 2013-03-24; First posted 2013-04-02 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Low Back Pain
Keywords: low back pain; Manual Therapy; Randomized Controlled Trial; Quality of life
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Craniosacral Therapy Program (Experimental): A program of 10 craniosacral therapy techniques
  Interventions: Other: Craniosacral Therapy Program
- One technique of craniosacral therapy (Active Comparator): Decompression L5-S1.
  Interventions: Other: One technique of craniosacral therapy

INTERVENTIONS:
Other: Craniosacral Therapy Program — The ten techniques of craniosacral therapy program are: Still Point (CV-4, Sacred Feet), diaphragms(pelvic, respiratory, thoracic inlet, hyoid, Occipital Cranial Base), Decompression L5-S1, Dural Tube Glide, Lift Front, Parietal Lift, Compression / decompression of the joint sphenobasilar, Temporary Technique, Compression / decompression of the temporomandibular joints, and Still Point CV-4.
  Arms: Craniosacral Therapy Program
Other: One technique of craniosacral therapy — Decompression L5-S1: lumbosacral decompression
  Arms: One technique of craniosacral therapy

SUMMARY:
The purpose of this study is to determine whether a craniosacral therapy program are effective on disability, quality of life, autonomic nervous system and oxidative stress indicators in patients with chronic low back pain.

DETAILED DESCRIPTION:
Design: Randomized clinical trial. Objective: to determine the effectiveness of a craniosacral therapy program on disability, quality of life, autonomic nervous system, body mass, hormonal indicators, spinal projection, and oxidative stress indicators in patients with chronic low back pain.

Participants: Seventy patients with chronic non-specific low back pain will be randomly assigned to an experimental and control group.

Intervention: For 10-week, the experimental group will undergo treatment comprising 10 sessions (1/week) of a craniosacral therapy program with ten techniques, and the control group will receive only one craniosacral technique.

Main Outcome Measures: disability, quality of life, biochemical estimation interstitial fluid, body mass indicators, hormonal indicators, indicators of autonomic nervous system,and indicators of oxidative stress will be collected in both groups at baseline, 10 weeks and 15 weeks after the last intervention in the experimental and control groups, by an assessor blinded to the treatment allocation of the patients. Baseline demographic and clinical variables will be examined between both groups with an independent Student t-test for continuous data. Separate 2x3 model ANOVA with time (baseline, 10 weeks and 15 weeks) as the within-subjects factor, group (experimental, control) will be to determine the effects of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain for > 3 months
* Score > 4 on the Roland Morris Disability questionnaire
* No undergoing another physical therapy treatment

Exclusion Criteria:

* Clinical signs of radiculopathy
* Presence of lumbar stenosis
* Fibromyalgia
* Spondylolisthesis
* History of spinal surgery
* Treatment with corticosteroids in the past two weeks
* Disease of the central or peripheral nervous system

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change for the Roland Morris Disability Questionnaire | At baseline, 10 weeks and 15 weeks
  The Roland Morris Disability Questionnaire is a self-administered disability measurement scored on a 24-point scale from 0 = no disability to 24 = severe disability

SECONDARY OUTCOMES:
Change for the Lifestyle indicators | At baseline, 10 weeks and 15 weeks
  Estimation interstitial fluid biochemistry and measure the following indicators: body mass, hormonal, autonomic nervous system and oxidative stress.
Change on Neural Network Analysis | At baseline, 10 weeks and 15 weeks
  Analysis of the projection on the spine and segmental innervation projection
Change on Quality of Life | At baseline, 10 weeks and 15 weeks
  SF-36 Health questionnaire scores range from 0 to 100% and indicate the self-perceived health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Adelaida Castro-Sánchez, PhD, Study Director — Universidad de Almeria
Locations (1):
- Universidad de Almeria, Almería, Almeria, Spain

REFERENCES:
- [Background] Arnadottir TS, Sigurdardottir AK. Is craniosacral therapy effective for migraine? Tested with HIT-6 Questionnaire. Complement Ther Clin Pract. 2013 Feb;19(1):11-4. doi: 10.1016/j.ctcp.2012.09.003. Epub 2012 Nov 9. PMID 23337558
- [Background] Jakel A, von Hauenschild P. A systematic review to evaluate the clinical benefits of craniosacral therapy. Complement Ther Med. 2012 Dec;20(6):456-65. doi: 10.1016/j.ctim.2012.07.009. Epub 2012 Aug 22. PMID 23131379
- [Background] Curtis P, Gaylord SA, Park J, Faurot KR, Coble R, Suchindran C, Coeytaux RR, Wilkinson L, Mann JD. Credibility of low-strength static magnet therapy as an attention control intervention for a randomized controlled study of CranioSacral therapy for migraine headaches. J Altern Complement Med. 2011 Aug;17(8):711-21. doi: 10.1089/acm.2010.0277. Epub 2011 Jul 6. PMID 21732734
- [Background] Harrison RE, Page JS. Multipractitioner Upledger CranioSacral Therapy: descriptive outcome study 2007-2008. J Altern Complement Med. 2011 Jan;17(1):13-7. doi: 10.1089/acm.2009.0644. Epub 2011 Jan 9. PMID 21214395
- [Background] Castro-Sanchez AM, Mataran-Penarrocha GA, Sanchez-Labraca N, Quesada-Rubio JM, Granero-Molina J, Moreno-Lorenzo C. A randomized controlled trial investigating the effects of craniosacral therapy on pain and heart rate variability in fibromyalgia patients. Clin Rehabil. 2011 Jan;25(1):25-35. doi: 10.1177/0269215510375909. Epub 2010 Aug 11. PMID 20702514
- [Background] Elden H, Ostgaard HC, Glantz A, Marciniak P, Linner AC, Olsen MF. Effects of craniosacral therapy as adjunct to standard treatment for pelvic girdle pain in pregnant women: a multicenter, single blind, randomized controlled trial. Acta Obstet Gynecol Scand. 2013 Jul;92(7):775-82. doi: 10.1111/aogs.12096. Epub 2013 Mar 4. PMID 23369067
- [Background] Gillespie BR. Case study in attention-deficit/hyperactivity disorder: the corrective aspect of craniosacral fascial therapy. Explore (NY). 2009 Sep-Oct;5(5):296-8. doi: 10.1016/j.explore.2009.06.003. No abstract available. PMID 19733816
- [Background] Mataran-Penarrocha GA, Castro-Sanchez AM, Garcia GC, Moreno-Lorenzo C, Carreno TP, Zafra MD. Influence of craniosacral therapy on anxiety, depression and quality of life in patients with fibromyalgia. Evid Based Complement Alternat Med. 2011;2011:178769. doi: 10.1093/ecam/nep125. Epub 2011 Jun 15. PMID 19729492
- [Background] Holla M, Ijland MM, van der Vliet AM, Edwards M, Verlaat CW. [Death of an infant following 'craniosacral' manipulation of the neck and spine]. Ned Tijdschr Geneeskd. 2009 Apr 25;153(17):828-31. Dutch. PMID 19469218
- [Background] Mann JD, Faurot KR, Wilkinson L, Curtis P, Coeytaux RR, Suchindran C, Gaylord SA. Craniosacral therapy for migraine: protocol development for an exploratory controlled clinical trial. BMC Complement Altern Med. 2008 Jun 9;8:28. doi: 10.1186/1472-6882-8-28. PMID 18541041
- [Background] Gerdner LA, Hart LK, Zimmerman MB. Craniosacral still point technique: exploring its effects in individuals with dementia. J Gerontol Nurs. 2008 Mar;34(3):36-45. doi: 10.3928/00989134-20080301-04. PMID 18350746
- [Background] McManus V, Gliksten M. The use of CranioSacral therapy in a physically impaired population in a disability service in southern Ireland. J Altern Complement Med. 2007 Nov;13(9):929-30. doi: 10.1089/acm.2007.0521. No abstract available. PMID 18047438
- [Background] Downey PA, Barbano T, Kapur-Wadhwa R, Sciote JJ, Siegel MI, Mooney MP. Craniosacral therapy: the effects of cranial manipulation on intracranial pressure and cranial bone movement. J Orthop Sports Phys Ther. 2006 Nov;36(11):845-53. doi: 10.2519/jospt.2006.36.11.845. PMID 17154138
- [Background] Flynn TW, Cleland JA, Schaible P. Craniosacral therapy and professional responsibility. J Orthop Sports Phys Ther. 2006 Nov;36(11):834-6. doi: 10.2519/jospt.2006.0112. No abstract available. PMID 17154136
- [Background] Bergkvist H. [A reflection over craniosacral therapy]. Ugeskr Laeger. 2005 Oct 3;167(40):3801-2. No abstract available. Danish. PMID 16221407
- [Background] Maher CG. Effective physical treatment for chronic low back pain. Orthop Clin North Am. 2004 Jan;35(1):57-64. doi: 10.1016/S0030-5898(03)00088-9. PMID 15062718
- [Background] Moran RW, Gibbons P. Intraexaminer and interexaminer reliability for palpation of the cranial rhythmic impulse at the head and sacrum. J Manipulative Physiol Ther. 2001 Mar-Apr;24(3):183-90. PMID 11313614
- [Background] Green C, Martin CW, Bassett K, Kazanjian A. A systematic review of craniosacral therapy: biological plausibility, assessment reliability and clinical effectiveness. Complement Ther Med. 1999 Dec;7(4):201-7. doi: 10.1016/s0965-2299(99)80002-8. PMID 10709302
- [Background] Upledger JE. Craniosacral therapy. Phys Ther. 1995 Apr;75(4):328-30. doi: 10.1093/ptj/75.4.328. No abstract available. PMID 7899490